CLINICAL TRIAL: NCT05183490
Title: Phase I Study of Adoptive Immunotherapy of Refractory Viral Infection with Ex Vivo Expanded Rapidly Generated Virus Specific T (R-MVST) Cells
Brief Title: R-MVST Cells for Treatment of Viral Infections
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Pawel Muranski, Assistant Professor of Medicine and Pathology and Cell Biology, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAS9079
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Epstein-Barr Virus Infections; Cytomegalovirus Infections; Adenovirus; BK Virus Infection
Keywords: Rapidly generated virus specific T cells (R-MVST); Refractory viral reactivation
MeSH Terms: conditions — Epstein-Barr Virus Infections; Cytomegalovirus Infections; Adenoviridae Infections | interventions — Cell Count

STUDY DESIGN:
Intervention Model Description: This is a single center, Phase 1, non-randomized open-label dose escalation study in two groups of immunocompromised patients. The recipients of allogeneic HCT who have will be enrolled in Group A, while SOT recipients will be enrolled in Group B. Each group will undergo independent dose escalation.
  Dose levels selected for Group A are based on previous experience with VST cells in HCT recipients and are lower than in Group B (SOT recipients), as donor-derived R-MVST cells are more likely to persist in recipients of HCT from the same donors. Thus, there is theoretically a higher risk for development of GVHD in this subset of patients. Starting dose proposed for Group B is based on our previous experience with virus-specific cells used for therapy of JC-PML, where multiple infusions of PyVST cells were used at the doses of up to 2x106 TNC/kg. R-MVST cells will target a particular virus (or several viruses), based on the pattern of viral reactivation seen in each patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Allogenic Stem Cell Transplant Recipient (SCT) (Experimental): Dose levels selected for Group A are based on previous experience with VST cells in HCT recipients and are lower than in Group B (SOT recipients), as donor-derived R-MVST cells are more likely to persist in recipients of HCT from the same donors. Thus, there is theoretically a higher risk for development of GVHD in this subset of patients. Each group will undergo independent dose escalation.
  Subjects will receive a single dose of R-MVST Cells, and followed for toxicity and GVHD for 28 days days after infusion. Up to two additional doses may be administered, minimum of 28 days apart if cohort safety is established and reinfusion criteria are met. A new 28-day safety-monitoring period will ensue for each additional infusion. Subjects will be followed for possible virological and clinical responses for up to 1 year after the initial R-MVST infusion.
  Interventions: Drug: Rapidly generated virus specific T (R-MVST) cells
- Group B: Solid organ transplant recipients (SOT) (Experimental): In SOT recipients, the study will use higher doses of R-MVST cells, as the infused anti-viral T cells are less likely to persist long-term and cause GVHD, based on the safety profile of PyVST cells used for therapy of PML in non-HCT subjects.
  Subjects will receive a single dose of R-MVST Cells, and followed for toxicity and GVHD for 28 days days after infusion. Up to two additional doses may be administered, minimum of 28 days apart if cohort safety is established and reinfusion criteria are met. A new 28-day safety-monitoring period will ensue for each additional infusion. Subjects will be followed for possible virological and clinical responses for up to 1 year after the initial R-MVST infusion.
  Interventions: Drug: Rapidly generated virus specific T (R-MVST) cells

INTERVENTIONS:
Drug: Rapidly generated virus specific T (R-MVST) cells — The R-MVST products will be manufactured individually for each patient from a selected donor; it is an anti-viral prophylaxis and treatment of viral reactivation.
  SCT dose escalation:
  Cohort / R-MVST dose
  * (-1A) 0.25x10^6 R-MVST TNC/kg
  * (1A) 0.5x10^6 R-MVST TNC/kg
  * (2A) 1x10^6 R-MVST TNC/kg
  SOT dose escalation:
  Cohort / R-MVST dose
  * (-1B) 1x10^6 R-MVST TNC/kg
  * (1B) 2x10^6 R-MVST TNC/kg
  * (2B) 4x10^6 R-MVST TNC/kg
  Other Names: R-MVST infusion

SUMMARY:
The primary objective is to determine the safety and feasibility of administering R-MVST cells to patients with refractory viral reactivation and/or symptomatic disease caused by Epstein Barr Virus (EBV), cytomegalovirus (CMV), adenovirus (ADV) or BK virus. R-MVST cells will be generated on-demand from the closest partially human leukocyte antigen (HLA)-matched (minimum haploidentical) healthy donors or from the original allo-transplant donor if available. The investigator will closely monitor the recipients for potential toxicities including graft-versus-host disease (GVHD) post-infusion.

Secondary objectives are to determine the effect of R-MVST infusion on viral load, possible recovery of antiviral immunity post-infusion and for evidence of clinical responses and overall survival. Recipients will be monitored for secondary graft failure at day 28 post R-MVST infusion.

DETAILED DESCRIPTION:
Starting from childhood, majority of healthy humans are exposed to common viruses such as CMV, EBV, BK and related human polyomaviruses and herpes viruses. Under normal circumstances those infections are well controlled by the adaptive immune system, but never eliminated. Instead, they are fairly inactive and produce relatively few consequences or symptoms. However, when T cell mediated immunity is suppressed, those dormant viruses reactivate and can cause a significant end-organ or severe systemic syndrome. This viral reactivation contributes to morbidity and mortality in recipients of allogeneic stem cell transplant (HCT) and solid organ transplants (SOT), and can affect many other patients who receive immunosuppressive therapies or have underlying pathology that affects T cell function, including patients with autoimmune diseases, congenital immunodeficiencies or HIV/AIDS. As a result of a weakened immune response, conventional antiviral prophylaxis or treatment with acyclovir and ganciclovir/foscarnet (for CMV) or rituximab (against EBV) are not always effective.

The main purpose of this study is to test whether giving an experimental cell product can treat the viral infection in patients who have conditions that cause poor function of their immune system, such as infections caused by viruses such as Cytomegalovirus (CMV), Epstein-Barr Virus (EBV), BK virus, or adenovirus. The cell product is called rapidly generated virus specific T cells or R-MVST.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Men and women ages 18 years or older of all ethnic groups will be eligible for the treatment
* Patients with history of HCT or SOT who demonstrate evidence of viral reactivation and/or infection manifesting as end-organ or systemic disease due to one or more of the following viruses: EBV, CMV, ADV or BK virus and suboptimal response to the standard of care therapy.
* Recurrent or Multiple Viral Infection. RVI defined as occurrence of more than one episode of reactivation that required intervention or symptomatic disease in recipient of allogeneic HCT that required standard of care treatment. MVI defined as more than one virus reactivating (defined by PCR positivity) or causing symptomatic systemic or end-organ disease. At least one of those viral reactivations required standard of care intervention. No standard of care therapy is defined for ADV and BK. Patients with multiple infections/reactivations will be eligible as long as at least one of those viral infections meet the criterium of "refractory".

Recipient Exclusion Criteria:

* Patients with other uncontrolled infections, except for CMV, EBV, ADV or BK. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to the day of infusion. For fungal infections, patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to R-MVST infusion. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection
* Patients who receive corticosteroids at ≥ 0.5mg/kg prednisone or equivalent.
* Patients who received anti-thymocyte globulin (ATG, Alemtuzumab (Campath), or other T-Cell immunosupressive monoclonal antibodies in the last 28 days.
* Patients who received methotrexate, or other antimetabolite-type immunosuppressants that are toxic to proliferating T cells in the last 7 days.
* Patients who received extracorporeal photopheresis within the last 28 days.
* Patients who received checkpoint inhibitor agents (e.g., nivolumab, pembrolizumab, ipilimumab) within 3 drug half-lives of the most recent dose to the infusion of R-MVST.
* Received donor lymphocyte infusion in last 28 days.
* Evidence of GVHD ≥ grade 2
* Evidence of biopsy-proven acute rejection in SOT recipients
* Active and uncontrolled relapse of malignancy
* Patients who are pregnant, or breastfeeding.
* Female of childbearing potential, or male with a female partner of childbearing potential, unwilling to use a highly effective method of contraception.
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who have received investigational (IND) product within 14 days of infusion of the the R-MVST cells.

Donor inclusion and exclusion criteria will be followed as per the most current BMT SOP (Donor selection, Donor evaluation and Donor Deferral).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity that leads to safety endpoint | Up to 28 days post R-MVST infusion
  This is to measure the incidence of toxicity post-infusion. Toxicities to consider include: GI toxicity, renal toxicity, hemorrhagic toxicity, cardiovascular toxicity hypotension, cardiac arrhythmia and left ventricular systolic dysfunction), neurological toxicity (somnolence and seizure), coagulation toxicity, vascular toxicity and pulmonary toxicity.
Incidence of GVHD post-infusion that leads to safety endpoint | Up to 28 days post R-MVST infusion
  This is to measure the incidence of GVHD post-infusion. The safety endpoint will be defined as de novo acute GVHD grade IV within 28 days of the last dose of R-MVST, or grades 3-5 infusion related adverse events within 28 days of the last CTL dose, or grades 4-5 non-hematological adverse events within 28 days of the last CTL dose that are not due to the pre-existing infection or the original malignancy or pre-existing co-morbidities as defined by the N a t i o n a l C a n c e r I n s t i t u t e ( NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.

SECONDARY OUTCOMES:
Percentage of subjects with good response in viral load or end-organ disease improvement | Up to 1 year after the initial R-MVST infusion
  This is to measure the effect of R-MVST infusion on viral load and possible recovery of antiviral immunity post-infusion. Subjects with complete response, partial response and stable disease will be tallied.
  If patient has end-organ involvement, the disease will be monitored for the evidence of clinical response. In case of PTLD/EBV lymphoma, the standard Cheson criteria will be applied (Cheson, Pfistner et al. 2007) for adult patients.
Overall survival rate | Up to 1 year after the initial R-MVST infusion
  This is to measure the effect of R-MVST infusion on viral load and possible recovery of antiviral immunity post-infusion. The percentage of people in a study or treatment group who are still alive for a certain period of time after they were diagnosed with or started treatment for a disease, such as cancer. The overall survival rate is often stated as a five-year survival rate, which is the percentage of people in a study or treatment group who are alive five years after their diagnosis or the start of treatment. Also called survival rate.
Incidence of secondary graft failure | Day 28 post R-MVST infusion
  Secondary graft failure is defined as initial neutrophil engraftment followed by subsequent decline in the ANC to < 500/mm3 for three consecutive measurements on different days, unresponsive to growth factor therapy that persists for at least 14 days in the absence of a known cause such as relapse. Secondary graft failure will be assessed at 28 days post R-MVST infusion in allo-HCT recipients and in recipients of solid organ transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Muranski, MD, Principal Investigator — Assistant Professor of Medicine and Pathology and Cell Biology
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Englund J, Feuchtinger T, Ljungman P. Viral infections in immunocompromised patients. Biol Blood Marrow Transplant. 2011 Jan;17(1 Suppl):S2-5. doi: 10.1016/j.bbmt.2010.11.008. No abstract available. PMID 21195305
- [Background] Tanaka Y, Kurosawa S, Tajima K, Tanaka T, Ito R, Inoue Y, Okinaka K, Inamoto Y, Fuji S, Kim SW, Tanosaki R, Yamashita T, Fukuda T. Analysis of non-relapse mortality and causes of death over 15 years following allogeneic hematopoietic stem cell transplantation. Bone Marrow Transplant. 2016 Apr;51(4):553-9. doi: 10.1038/bmt.2015.330. Epub 2016 Jan 11. PMID 26752142
- [Background] Hill JA, Mayer BT, Xie H, Leisenring WM, Huang ML, Stevens-Ayers T, Milano F, Delaney C, Sorror ML, Sandmaier BM, Nichols G, Zerr DM, Jerome KR, Schiffer JT, Boeckh M. The cumulative burden of double-stranded DNA virus detection after allogeneic HCT is associated with increased mortality. Blood. 2017 Apr 20;129(16):2316-2325. doi: 10.1182/blood-2016-10-748426. Epub 2017 Feb 16. PMID 28209721